CLINICAL TRIAL: NCT02468752
Title: Mängden kvävgasbubblor i Blodet Efter Dykning Vid Syrgasandning jämfört Med Luftandning
Brief Title: Reduction of Venous Emboli Load After Breathing Normobaric Oxygen Compared to Air
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Swedish Armed Forces Diving and Naval Medicine Centre (Other); KTH Royal Institute of Technology (Other); Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Nicklas Oscarsson, MD, Göteborg University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: DYK 14-16
Record Dates: First submitted 2015-06-03; First posted 2015-06-11 (Estimated); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Hyperbaric; Diving Medicine; Decompression Sickness; Central Nervous Injury; Inflammation; Endothelial Dysfunction
MeSH Terms: conditions — Decompression Sickness; Inflammation | interventions — Oxygen; Air

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Air (Sham Comparator): Normobaric air breathing
  Interventions: Other: Air
- Oxygen (Experimental): Normobaric oxygen breathing
  Interventions: Drug: Oxygen

INTERVENTIONS:
Drug: Oxygen
  Arms: Oxygen
Other: Air
  Arms: Air

SUMMARY:
Primary objective:

- Assessment of venous gas emboli load post diving when breathing normobaric oxygen compared to air.

Secondary objective:

* Assessment of fluid markers of central nervous system injury in blood post diving
* Assessment of fluid markers of inflammation and endothelial dysfunction in blood post diving

Tertiary objective:

- Assessment of DCS frequency

DETAILED DESCRIPTION:
This is a prospective, double blinded, randomized, cross-over study in Sweden. The study was performed in two different sets, each containing standardized dives in a wet hyperbaric chamber. The dives included movement on depth.

In each study set 16-32 professional divers performed no-decompression dives to a depth of 42 metres of seawater (msw). The gas used during the dives was compressed air.

After surfacing the divers breathed either normobaric oxygen or normobaric air on a demand mask. Timing of oxygen/air-breathing differed between study sets. The content of breathing gas was unknown to both divers and examining personnel.

Immediately post dive the divers were assessed using either transthoracic doppler ultrasound (TTD) or transthoracic 2-D ultrasound (TTE) to determine VGE load, time to VGE detection and VGE duration.

Signs of DCS were actively sought.

TTD measurements were done every five minutes during the first 30 minutes, thereafter every 15 minutes during 90 minutes.

TTE was performed every 30 minutes, using an apical 4-chamber view.

Blood samples were obtained pre-dive, 30-45 minutes post-dive and 120 minutes post-dive.

Set 1: 16 divers, divided into two equal groups (A and B). Dive to 42 msw during 10 min with a safety stop at five msw during three min. Immediately post dive breathing of oxygen (group A) or air (group B) during 30 min. VGE load, time to VGE detection and VGE duration is recorded. Blood samples were obtained pre-dive and 30 and 120 minutes post-dive. After 48 hours, the dives were repeated with switched gases between the groups.

Set 2: 32 divers, divided into two equal groups (A and B). Dive to 42 msw during 10 min with a safety stop at five msw during three min. Fifteen minutes post dive breathing of oxygen (group A) or air (group B) during 30 min. VGE load, time to VGE detection and VGE duration is recorded. Blood samples were obtained pre-dive and 45 and 120 minutes post-dive, from the first 16 divers. After 48 hours, the dives were repeated with switched gases between the groups.

Two further planned sets with repeated diving and shorter duration of oxygen/air-breathing were never carried through.

AE including SAE will be recorded during the study. DCS may be considered either an AE or SAE depending on severity. Ongoing AE and SAE will be followed up.

ELIGIBILITY:
Inclusion Criteria:

* Professional diver
* Fit to dive according to Swedish Navy standards

Exclusion Criteria:

* NONE

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Venous gas emboli | 120 minutes
  Kisman-Masurel grading

SECONDARY OUTCOMES:
Inflammatory activity and endothelial dysfunction | 120 minutes/ 48 hours
  E.g. VCAM-1, ICAM-1
Decompression sickness | 24 hours
  Clinical diagnosis
Markers of central nervous system injury | 120 minutes/ 48 hours
  E.g. GFAP, Tau, NfL, UCHL-1

CONTACTS AND LOCATIONS:
Overall Officials: Mikael Gennser, PhD, Principal Investigator — Kungliga Tekniska Högskolan, Stockholm, Sweden
Locations (2):
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Kungliga Tekniska Högskolan, Stockholm

IPD SHARING:
Plan to Share IPD: No